CLINICAL TRIAL: NCT04032769
Title: MOdified DIagnostic strateGy to Safely ruLe-out Pulmonary Embolism In the Emergency depArtment: A Non-Inferiority Cluster Cross-over Randomized Trial
Brief Title: Modified Strategy to Safely Rule Out Pulmonary Embolism in the Emergency Department
Acronym: MODIGLIA-NI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP180595
Record Dates: First submitted 2019-07-18; First posted 2019-07-25 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Pulmonary Embolism
Keywords: Pulmonary embolism; PERC Rule; Years Rule; Peps Rule; Emergency department
MeSH Terms: conditions — Pulmonary Embolism; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified strategy MODS (Experimental): the threshold of D-dimer will depend on the YEARS rule (MODS strategy):
  1. If all the three items of YEARS are negative (i.e. No hemoptysis, No clinical sign of deep venous thrombosis and PE is not the most likely diagnosis), then the threshold of D-dimer will be raised at 1000 ng/ml.
  2. If at least one item of YEARS is positive, then the threshold will remain unchanged (">500 ng/ml" for patients aged < 50 and "> agex10" for patients aged 50 and over).
     * A positive result of D-dimer and the absence of other obvious cause for PE will mandate a CTPA, or V/Q scan if CTPA is contra-indicated.
     * A negative result of D-dimer will rule out PE.
  Interventions: Other: MODS (MOdified Diagnostic Strategy)
- Control group (No Intervention): All included patients will be tested with D-Dimer, threshold for ordering a CTPA as usual

INTERVENTIONS:
Other: MODS (MOdified Diagnostic Strategy) — Modified diagnostic strategy (MODS):
  All included patients will be tested with quantitative D-dimer. The MODS work-up strategy will be based on YEARS rule, that included three criteria (hemoptysis, signs of DVT, PE is the most likely diagnosis)
  - If all YEARS criteria are absent, the threshold of D-Dimer for ordering a CTPA will be raised at 1000 ng/ml.
  If at least one criterion of YEARS is present, then the D-dimer threshold for ordering a CTPA will be as usual (500 ng/ml, or agex10 for patients aged 50 and over)
  Arms: Modified strategy MODS

SUMMARY:
Because a missed PE could be potentially lethal, several researches reported that PE is both overinvestigated and overdiagnosed. The diagnostic gold standard for PE is the computed tomographic pulmonary angiogram (CTPA) and has been shown to have clear risks and other downsides. To limit the use of CTPA, two rules were recently reported to be safe to exclude PE: the PERC rule and the YEARS rule. PERC is an 8 item block of clinical criteria that has recently been validated to safely exclude PE in low risk patients. YEARS is a clinical rule that allow to raise the threshold of D-dimer for the order of CTPA. However, whether a modified diagnostic algorithm that includes these two rules combined could safely reduce imaging study use in the ED is unknown.

This is a non-inferiority, cluster cross-over randomized, international trial.

Each center will be randomized on the sequence of period intervention: 4 months intervention (MOdified Diagnostic Strategy: MODS) followed by 4 months control (usual care), or 4 months control followed by 4 months intervention with 1 month of "wash-out" between the two periods.

All centers will recruit adult emergency patients with a suspicion of PE.

In the control group (usual strategy), patients will be tested for D-dimer, followed if positive by a CTPA.

In the intervention group (MODS) :

All included patients will be tested with quantitative D-dimer. The MODS work-up will be based on YEARS rule :

- If all YEARS criteria are absent, the threshold of D-Dimer for ordering a CTPA will be raised.

If at least one criterion of YEARS is present, then the D-dimer threshold for ordering a CTPA will be as usual.

DETAILED DESCRIPTION:
The diagnosis of Pulmonary Embolism (PE) is a crucial matter in the Emergency Department (ED). Because a missed PE could be potentially lethal, several researches reported that PE is both overinvestigated and overdiagnosed. The diagnostic gold standard for PE is the computed tomographic pulmonary angiogram (CTPA) and has been shown to have clear risks (allergic reaction, acute renal failure, delayed solid tumor) and other downsides such as prolonged ED stay and increased cost. To limit the use of CTPA, two rules were recently reported to be safe to exclude PE: the PERC rule and the YEARS rule.

PERC is an 8 item block of clinical criteria that has recently been validated to safely exclude PE in low risk patients.

YEARS is a clinical rule that allow to raise the threshold of D-dimer for the order of CTPA. However, whether a modified diagnostic algorithm that includes these two rules combined could safely reduce imaging study use in the ED is unknown.

The primary objective of this trial is to assess the safety of a modified diagnostic strategy (MODS) with the YEARS for patients in whom PE was not excluded by PERC score in the ED.

The primary endpoint is the failure percentage of the diagnostic strategy, defined as a diagnosed thrombo-embolic event at 3 month follow-up (either a PE or a deep venous thrombosis), among patients in whom PE has been initially ruled out.

The secondary outcomes try to assess the efficacy of the modified diagnostic strategy (MODS) in reducing order of irradiative imaging studies, ED length of stay, undue onset of anticoagulation regimen, hospital admission, hospital readmission, and mortality at 3 months.

To evaluate the efficacy of the modified diagnostic strategy to reduce overall 3-months total cost.

Secondary endpoints include:

* CTPA or V/Q scan
* Anticoagulant therapy administration
* Length of stay in the ED (hours)
* Admission to the hospital following ED visit.
* All causes re hospitalization at 3 months,
* Death from all causes at 3 months
* Diagnosed pulmonary embolism at 3 month follow-up excluding the isolated sub-segmental pulmonary embolism, among patients in whom PE has been initially ruled out
* PEPS score
* 3 months total cost and cost effectiveness

In the Modified diagnostic strategy (MODS), All included patients will be tested with quantitative D-dimer. The MODS work-up strategy will be based on YEARS rule, that included three criteria (hemoptysis, signs of DVT, PE is the most likely diagnosis)

- If all YEARS criteria are absent, the threshold of D-Dimer for ordering a CTPA will be raised at 1000 ng/ml.

If at least one criterion of YEARS is present, then the D-dimer threshold for ordering a CTPA will be as usual (500 ng/ml, or agex10 for patients aged 50 and over)

Group control :

All included patients will be tested with D-Dimer, the threshold for ordering a CTPA will be as usual (conventional age-adjusted threshold at 500 ng/ml, or agex10 for patients aged 50 and over).

Safely reducing the use of CTPA would be beneficial for the patients, by limiting their risk of associated adverse events and overdiagnosis of PE, and will also reduce their length of stay in the ED, which is associated with better outcomes. Furthermore, reducing supplemental investigations for patients with suspicion of PE may also reduce the cost of ED visits, which would be of great benefit in the context of increasingly resource stretched healthcare services.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged ≥ 18 years that presents to an ED
* With new onset of or worsening of shortness of breath or chest pain or syncope

Exclusion Criteria:

* Opposition to the participation to the study
* Anticipated inability to follow up at 3 month
* Other obvious cause than PE for chest pain, syncope or dyspnea
* High clinical probability of PE (estimated by the physician gestalt as > 50%) or low clinical probability and PERC negative patients
* Low clinical probability (estimated by the physician gestalt as < 15%) and no item of the PERC score (heart rate > 100, Sa02 < 95, unilateral leg swelling, hemoptysis, past history of thrombo-embolism, exogen estrogen intake, recent trauma or surgery, age ≥ 50)
* Acute severe presentation (clinical signs of respiratory distress, hypotension, SpO2<90%, shock)
* Concurrent anticoagulation treatment
* Current diagnosed thrombo-embolic event (in the past 6 months)
* Prisoners
* Pregnancy
* No social security
* Participation in another intervention trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1414 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2020-11-20 (Actual)

PRIMARY OUTCOMES:
the failure percentage of the diagnostic strategy, defined as a diagnosed thrombo-embolic event at 3 month follow-up | 3 months follow up
  existence of a diagnosed thrombo embolic event (PE or DVT) among patients in whom PE has been initially ruled out.

SECONDARY OUTCOMES:
reduced irradiative imaging studies | 3 months follow up
  CTPA or V/Q scan
ED length of stay | Through ED Discharge within 24 hours
  length of stay in the ED (hours)
anticoagulant therapy administration | 3 months follow up
  onset of anticoagulant regimen
hospital admission | 3 months follow up
  admission to the hospital following ED visit
hospital re admission | 3 months
  all causes re hospitalization at 3 months
mortality | 3 months
  Death from all causes at 3 months
Safety of the PEPS score | 3 months
  performance characteristic of the PEPS score for the diagnosis of PE both in the ED and at 3 Months. The false negative rate of PEPS score will be tested, as the theoretical percentage of indicated CTPA according to its value.
total cost and cost effectiveness | 3 months
  total cost and cost effectiveness (cost per major adverse event averted, namely hospitalisation, rehospitalisation, imaging study, death).

CONTACTS AND LOCATIONS:
Overall Officials: Yonathan Freund, professor, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (2):
- Emergency department Hospital Pitié-Salpêtrière, Paris, France
- Emergency department, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Yes, upon request, after approval by the primary investigator and clinical research platform of East Paris. For the purpose of IPD meta-analysis, or secondary analysis. Unidentifying data will be shared.

REFERENCES:
- [Derived] Nze Ossima A, Ngaleu Siaha BF, Mimouni M, Mezaour N, Darlington M, Berard L, Cachanado M, Simon T, Freund Y, Durand-Zaleski I. Cost-effectiveness of modified diagnostic strategy to safely rule-out pulmonary embolism in the emergency department: a non-inferiority cluster crossover randomized trial (MODIGLIA-NI). BMC Emerg Med. 2023 Nov 29;23(1):140. doi: 10.1186/s12873-023-00910-x. PMID 38030975
- [Derived] Freund Y, Chauvin A, Jimenez S, Philippon AL, Curac S, Femy F, Gorlicki J, Chouihed T, Goulet H, Montassier E, Dumont M, Lozano Polo L, Le Borgne P, Khellaf M, Bouzid D, Raynal PA, Abdessaied N, Laribi S, Guenezan J, Ganansia O, Bloom B, Miro O, Cachanado M, Simon T. Effect of a Diagnostic Strategy Using an Elevated and Age-Adjusted D-Dimer Threshold on Thromboembolic Events in Emergency Department Patients With Suspected Pulmonary Embolism: A Randomized Clinical Trial. JAMA. 2021 Dec 7;326(21):2141-2149. doi: 10.1001/jama.2021.20750. PMID 34874418
- [Derived] Philippon AL, Dumont M, Jimenez S, Salhi S, Cachanado M, Durand-Zaleski I, Simon T, Freund Y. MOdified DIagnostic strateGy to safely ruLe-out pulmonary embolism In the emergency depArtment: study protocol for the Non-Inferiority MODIGLIANI cluster cross-over randomized trial. Trials. 2020 Jun 3;21(1):458. doi: 10.1186/s13063-020-04379-y. PMID 32493383